CLINICAL TRIAL: NCT02775669
Title: Non-invasive Epicutaneous Transfontanel Intracranial Pressure Monitoring in Children Under the Age of One: a Novel Technique
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Clinic Frankfurt (Other)
Responsible Party: Principal Investigator, Bedjan Behmanesh, MD, University Clinic Frankfurt
Other Study IDs: 34/15
Record Dates: First submitted 2016-05-10; First posted 2016-05-17 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Hydrocephalus
Keywords: noninvasive ICP monitoring
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- intracranial ICP monitoring: invasive intracranial ICP monitoring
- tranfontanel ICP monitoring: Noninvasive transfontanel ICP monitoring

SUMMARY:
Investigators compare the ICP of two standard Spiegelberg ICP-probes in children, which underwent an operation due to craniosynostosis.

DETAILED DESCRIPTION:
The investigators compare the ICP of two standard Spiegelberg ICP-probes in children, which underwent an operation and Implantation of an external ventricle drain or a subdural ICP Monitoring devise. The second ICP probe is fixed epicutaneously on the skin over the frontal fontanel. The hourly measured ICPs within 24 hours postoperatively were compared with the Bland-Altman two methods analysis.

ELIGIBILITY:
Inclusion Criteria:

Child with open fontanel Need of ICP monitoring

Exclusion Criteria:

closed fontanel No Need of ICP monitoring

Ages: 1 Day to 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study Population: Children with open fontanels and need of intracranial pressure monitoring
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of ICP values (mmHg), intracranial pressure obtained invasive and noninvasive in mmHg will be compared. Either there is a significant difference or not. The data will be collected hourly. Device: Spiegelberg ICP Probe. | 24 hours
  ICP values in mmHg will be collected in both arms